CLINICAL TRIAL: NCT03374306
Title: Treatment Effect of Topical Application of Low-concentration (0.01%) Atropine on the Human Eye With Fast and Slow Myopia Progression Rate as Classified by Electro-retinal Responses
Brief Title: Topical Application of Low-concentration (0.01%) Atropine on the Human Eye With Fast and Slow Myopia Progression Rate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Henry HL Chan, PhD, Association Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HongKongPU_Optometry1
Record Dates: First submitted 2017-12-11; First posted 2017-12-15 (Actual); Results first posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Myopia
Keywords: Myopia; Myopia control; Atropine; Electroretinogram; Multifocal Electroretinogram
MeSH Terms: conditions — Myopia | interventions — Atropine; Lubricant Eye Drops

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Who Masked: Participant, Investigator
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Atropine 0.01% (Experimental): Group receiving atropine treatment for 18 months
  Interventions: Drug: Atropine (0.01%)
- Artifical tear (Placebo Comparator): Group receiving placebo for 18 months
  Interventions: Drug: Artificial tear

INTERVENTIONS:
Drug: Atropine (0.01%) — tropical application
  Arms: Atropine 0.01%
Drug: Artificial tear — tropical application
  Arms: Artifical tear

SUMMARY:
Our project is a 24-month longitudinal randomized controlled trial that aims to investigate the myopia development after topical application of 0.01% atropine in children with either fast or slow myopia progression classified according to their initial electro-retinal responses. This will help elucidate the effectiveness of using low concentration atropine for myopia control in children with different myopia progression rates.

ELIGIBILITY:
Inclusion Criteria:

* Age between 7 and 10 years
* Good general health and no family history of ocular diseases
* No current or history of epilepsy or asthma
* Myopia : -0.50 to -1.00 D (inclusive, both eyes)
* Astigmatism : ≤ 0.50 D
* No hyperopia, amblyopia or strabismus
* No reported ocular eye diseases or disorders
* No drug allergy

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 71 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry HL CHAN, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- School of Optometry, Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: Feb 2018 - Oct 2018 Location: HK PolyU Optometry clinic
Period: Overall Study
Arm/Group | Atropine 0.01% | Artifical Tear
Started | 36 | 35
Completed | 34 | 27
Not Completed | 2 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Atropine 0.01% | Artifical Tear | Total
Number analyzed (Participants) | 36 | 35 | 71
Age, Categorical [Count of Participants; unit: Participants] — Population: 2 subjects from treatment group and 8 subjects from control group withdrew from the study
  Participants
    number analyzed (Participants) | 34 | 27 | 61
    <=18 years | 34 | 27 | 61
    Between 18 and 65 years | 0 | 0 | 0
    >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 2 subjects from treatment group and 8 subjects from control group withdrew from the study
  Participants
    number analyzed (Participants) | 34 | 27 | 61
    Female | 17 | 13 | 30
    Male | 17 | 14 | 31
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants] — Population: 2 subjects from treatment group and 8 subjects from control group withdrew from the study
  participants
    Hong Kong: number analyzed (Participants) | 34 | 27 | 61
    Hong Kong | 34 | 27 | 61
Refractive errors [Mean (Standard Deviation); unit: Dioptre] — Population: 2 subjects from treatment group and 8 subjects from control group withdrew from the study
  Dioptre
    number analyzed (Participants) | 34 | 27 | 61
    (all) | -1.88 (1.08) | -1.74 (0.71) | -1.8 (0.95)
Electroretinogram [Mean (Standard Deviation); unit: nV/deg^2] — Induced response from central retina measured by multifocal electroretinogram Population: 2 subjects from treatment group and 8 subjects from control group withdrew from the study
  nV/deg^2
    number analyzed (Participants) | 34 | 27 | 61
    (all) | 41.65 (24.4) | 50.01 (27.75) | 45.16 (25.45)
Axial length [Mean (Standard Deviation); unit: mm] — Population: 2 subjects from treatment group and 8 subjects from control group withdrew from the study
  mm
    number analyzed (Participants) | 34 | 27 | 61
    (all) | 24.17 (0.79) | 24.09 (0.74) | 24.13 (0.76)

OUTCOME MEASURES:

1. Primary Outcome: Annualized Changes in Refractive Error (SER)
Description: Annualized changes in refractive error (SER) after receiving the 0.01 atropine or artificial tears up to 18 months
Time Frame: 18 months
Population: Annualized changes in refractive error (SER)
Measure: Mean (Standard Deviation); unit: Dioptre/year
Arm/Group | Atropine 0.01% | Artifical Tear
Number analyzed (Participants) | 34 | 27
Dioptre/year | -0.70 (0.39) | -0.66 (0.41)

2. Secondary Outcome: Annualized Change in Axial Length
Description: Annualized change in axial length after receiving the 0.01 atropine or artificial tears up to 18 months
Time Frame: 18 months
Population: annualized change in axial length
Measure: Mean (Standard Deviation); unit: mm/year
Arm/Group | Atropine 0.01% | Artifical Tear
Number analyzed (Participants) | 34 | 27
mm/year | 0.3 (0.22) | 0.32 (0.16)

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Atropine 0.01% | Artifical Tear
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/27
Other Adverse Events (participants affected / at risk) | 0/34 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2018-01-01): https://cdn.clinicaltrials.gov/large-docs/06/NCT03374306/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-01): https://cdn.clinicaltrials.gov/large-docs/06/NCT03374306/SAP_001.pdf
  • Informed Consent Form (2018-02-02): https://cdn.clinicaltrials.gov/large-docs/06/NCT03374306/ICF_002.pdf